CLINICAL TRIAL: NCT06288295
Title: Retrospective Study on Data Aiming to Establish a Prediction Score for Return Home at the Time of Admission to a Multidisciplinary Medical Department
Brief Title: Retrospective Study on Data Aiming to Establish a Prediction Score for Return Home at the Time of Admission to a Multidisciplinary Medical Department (SCORDOM
Acronym: SCORDOM
Status: Completed | Type: Observational
Sponsor: Elsan (Other)
Responsible Party: Sponsor
Other Study IDs: Etude SCORDOM
Record Dates: First submitted 2024-02-09; First posted 2024-03-01 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Continuity of Patient Care
Keywords: predictive score; return to home; elderly

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Score development cohort: Patients over 60 years of age admitted to a general medicine department in the investigating center between October 2021 and February 2022
- Score validation cohort: Patients over 60 years of age admitted to a general medicine department in the investigating center between October 2022 and February 2023

SUMMARY:
The goal of this observational study is to define clinical, biological and socio-cultural criteria, from the very first days of hospitalization on the multidisciplinary medicine department, to guide the patient's discharge from hospital (return to home when discharged from hospital).

The data collected will be those contained in the medical records of patients over 60 years of age who were admitted to the multidisciplinary medical department between October 2021 and February 2022 and between October 2022 and February 2023.

This study also aims at developing and validating a predictive score of orientation at the end of hospitalisation.

Participants are patients previously hospitalized. They will be informed about the study by post and will be able to object to the use of his or her data.

ELIGIBILITY:
Inclusion Criteria:

For the development of the score:

1. All patients over 60 years of age admitted to the multidisciplinary medical department in the investigating center between October 2021 and February 2022.
2. Patients for whom data of interest to this study are available in medical records.

For score validation :

1. All patients aged over 60 admitted to the multidisciplinary medicine department of the investigating center between October 2022 and February 2023.
2. Patients for whom data of interest to this study are available in medical records.

Exclusion Criteria:

1. Patients transferred from an intensive care or continuing care unit
2. Patients in palliative care
3. Patients residing in an EHPAD (establishment for the elderly) or nursing home prior to hospitalization
4. Patients without a minimum blood test on admission (blood test less than 48 hours old)
5. Patients whose reason for hospitalization is due to COVID
6. Patients who have objected to the use of their personal data

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over 60 years of age, hospitalized in Nancy private Hospital Lorraine, in the multidisciplinary medical department, between october 2021 and February 2022, and patients hospitalized between October 2022 and February 2023 (in the same department).
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Number of patients with a return to home after hospitalization and with similar clinical parameters, similar age category, similar pathology and similar biological parameters | Hospital stay, up to 3 weeks
  Data collected among hospital data from october 2021 to february 2022. Clinical parameters measured: age, confusional syndrome, fever, eschar, blood pressure, etc; biological paremeters: (blood test performed in the last 2 days before discharge: albuminemia, natremia, protein C, Creatinemy, hemoglobinemy)

SECONDARY OUTCOMES:
Number of patients with a return to home after hospitalization and with similar clinical parameters, similar age category, similar pathology and similar biological parameters | Hospital stay, up to 3 weeks
  Data collected among hospital data from october 2022 to february 2023. Clinical parameters measured: age, confusional syndrome, fever, eschar, blood pressure, etc; biological paremeters: (blood test performed in the last 2 days before discharge: albuminemia, natremia, protein C, Creatinemy, hemoglobinemy)

CONTACTS AND LOCATIONS:
Overall Officials: Anais Bauer, PhD, Principal Investigator — Hôpital Privé Nancy Lorraine
Locations (1):
- Hôpital Privé Nancy Lorraine, Nancy, France